CLINICAL TRIAL: NCT07222566
Title: AN INTERVENTIONAL PHASE 3, DOUBLE-BLIND, RANDOMIZED STUDY TO EVALUATE EFFICACY AND SAFETY OF PF-08634404 IN COMBINATION WITH CHEMOTHERAPY VERSUS PEMBROLIZUMAB IN COMBINATION WITH CHEMOTHERAPY IN ADULT PARTICIPANTS WITH LOCALLY ADVANCED OR METASTATIC NON-SMALL CELL LUNG CANCER
Brief Title: A Study to Learn About the Study Medicine Called PF-08634404 in Combination With Chemotherapy in Adult Participants With Locally Advanced or Metastatic Non-Small Cell Lung Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C6461001; 2025-523461-17-00 (Registry Identifier: CTIS (EU)); Symbiotic-Lung-01 (Other: Pfizer)
Record Dates: First submitted 2025-10-28; First posted 2025-10-30 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Advanced Non-Small Cell Lung Cancer; Non-Small Cell Lung Cancer; Carcinoma, Non-Small-Cell Lung; Carcinoma, Non-Small-Cell Lung (NSCLC); Metastatic Non Small Cell Lung Cancer; Lung Cancer
Keywords: non-squamous NSCLC; squamous NSCLC; metastatic (Stage IV) squamous or non-squamous NSCLC; Advanced or Metastatic Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Carcinoma; Lung Neoplasms; Neoplasm Metastasis | interventions — pembrolizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: This is double-blind study, neither the participants nor the study team will know whether the participants are receiving PF-08634404 or Pembrolizumab.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Arm A (Experimental): Participants will receive PF-08634404 combined with chemotherapy regimen 1, followed by maintenance therapy with PF-08634404.
  Interventions: Biological: PF-08634404; Drug: Chemotherapy Regimen 1
- Arm B (Active Comparator): Participants will receive pembrolizumab combined with chemotherapy regimen 1, followed by maintenance therapy with pembrolizumab.
  Interventions: Biological: Pembrolizumab; Drug: Chemotherapy Regimen 1
- Arm C (Experimental): Participants will receive PF-08634404 combined with chemotherapy regimen 2, followed by maintenance therapy with PF-08634404 and chemotherapy.
  Interventions: Biological: PF-08634404; Drug: Chemotherapy Regimen 2
- Arm D (Active Comparator): Participants will receive pembrolizumab combined with chemotherapy regimen 2, followed by maintenance therapy with pembrolizumab and chemotherapy.
  Interventions: Biological: Pembrolizumab; Drug: Chemotherapy Regimen 2

INTERVENTIONS:
Biological: PF-08634404 — Solution for infusion
  Arms: Arm A; Arm C
Biological: Pembrolizumab — Injection for IV use
  Arms: Arm B; Arm D
Drug: Chemotherapy Regimen 1 — Injection for IV use
  Arms: Arm A; Arm B
Drug: Chemotherapy Regimen 2 — Injection for IV use
  Arms: Arm C; Arm D

SUMMARY:
This study is being done to find out if a new medicine called PF-08634404, when given with chemotherapy, works better than the present standard treatment (pembrolizumab with chemotherapy) for adults with a type of lung cancer called non-small cell lung cancer (NSCLC) that is either locally advanced (spread to nearby tissues) or has spread to other parts of the body.

To join the study, participants must meet the following conditions:

* Be 18 years or older.
* Have locally advanced (Stage IIIB/IIIC) or metastatic (Stage IV) squamous or non-squamous NSCLC.
* Is not a candidate for complete surgical resection or curative chemoradiotherapy.
* Do not have known actionable genomic alterations
* Be treatment naïve for advanced or metastatic disease

Participants in this study will be assigned to two different parts of the study depending on their type of tumor: participants with squamous NSCLC will be assigned to Part 1, while participants with non-squamous NSCLC will be assigned to Part 2.

Each participant will be randomly assigned (like a flip of the coin) to one of two treatment groups in a blinded fashion:

* Part 1 - Arm A or Part 2 - Arm C (Experimental Group): Will receive a new study medicine called PF-08634404 along with a kind of chemotherapy specific to the type of tumor.
* Part 1 - Arm B or Part 2 - Arm D (Control Group): Will receive an approved medicine called pembrolizumab along with a kind of chemotherapy specific to the type of tumor.

Participants will receive their assigned treatment through intravenous (IV) infusions, which means the medicine is given directly into a vein. The treatment will be given in cycles, participants will receive PF-08634404 or Pembrolizumab in combination with chemotherapy followed by maintenance with either PF-08634404 or Pembrolizumab monotherapy (Part 1) or PF-08634404 or Pembrolizumab in combination with a chemotherapeutic drug (Part 2). Participants will continue receiving treatment if it is helping and not experiencing serious side effects.

The study will include regular visits for:

* Treatment and health checks: while participant continues receiving treatment.
* Tests to monitor how cancer responds: every 6 weeks during the first 48 weeks, then every 12 weeks thereafter.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older at screening.
* Have pathologically confirmed locally advanced (Stage IIIB/IIIC) or metastatic (Stage IV)squamous or non-squamous NSCLC and not be a candidate for complete surgical resection and curative concurrent/sequential chemoradiotherapy (according to the 9th edition of the Union for International Cancer Control and American Joint Committee on Cancer lung cancer Tumor, lymph nodes, metastasis (TNM) staging system).
* Have tumor tissue available, either paraffin block or slides from a core, excisional or fine needle biopsy
* PD-L1 status available based on local testing results
* Measurable disease based on RECIST v1.1 per investigator.
* Eastern Cooperative Oncology Group performance status (ECOG) score of 0 or 1
* Expected survival ≥12 weeks

Exclusion Criteria:

* Participants with known actionable genomic alteration (AGAs), including estimated glomerular filtration rate (EGFR), anaplastic lymphoma kinase (ALK), Repressor of Silencing 1 (ROS1), neurotrophic tyrosine receptor kinase (NTRK), v-raf murine sarcoma viral oncogene homolog B1 (BRAF), rearranged during transfection (RET), and mesenchymal-epithelial transition (MET), for which there are available first-line therapies per local standard-of-care (SOC) are ineligible. Documented negative results for EGFR, ALK, and ROS1 AGAs are required for participants with non-squamous histology.
* Known active CNS lesions are excluded. Participants with definitively treated brain metastases (surgery and/or radiotherapy) may be eligible. Clinically inactive brain metastases of longest diameter < 1 cm are permitted.
* Participants with clinically significant risk of hemorrhage or fistula are excluded.
* Participants with any history of another malignancy within 3 years before the first dose of study intervention, or any evidence of residual disease from a previously diagnosed malignancy.
* Unresolved toxicities from prior anti-tumor therapy, that did not recover to NCI CTCAE v5.0 Grade 0 or 1.
* Known to have a history of a severe allergy to any component of the study intervention, or a history of severe allergic reaction to chimeric or humanized antibody.
* History of allogeneic organ / hematopoietic stem cell transplantation.
* Participants with any of the following respiratory conditions:
* Evidence of noninfectious or drug-induced interstitial lung disease (ILD) or pneumonitis
* Grade ≥3 pulmonary disease unrelated to underlying malignancy
* History of uncontrolled comorbidities within 6 months prior to the first dose including uncontrolled cardiac and cerebrovascular conditions, hypertension, diabetes, significant vascular disease or arterial/severe venous thromboembolic events.
* Major surgery < 4 weeks or minor surgery < 3 days prior to first dose of study intervention.
* History of severe bleeding tendency or coagulation dysfunction
* History of esophageal varices, severe ulcers, unhealed wounds, gastrointestinal perforation, abdominal fistula, gastrointestinal obstruction, intra-abdominal abscess, or acute gastrointestinal bleeding within 6 months prior to the first dose.
* Participants with acute, chronic or symptomatic infections including participants positive for active HIV, hepatitis B virus (HBV), or Hepatitis C virus (HCV).
* Participants with history of immunodeficiency
* Any medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior (in the past 5 years) or laboratory abnormality that may increase the risk of study participation or make the participant inappropriate for the study.
* Previous systemic anti-tumor therapy including:

  1. Prior systemic therapy, including anti-PD-(L)1 therapy, for locally advanced, unresectable, or metastatic NSCLC.
  2. Previous treatment with immunotherapy
  3. Prior radiotherapy > 30 Gy to the lung < 6 months of first dose of study intervention
  4. Palliative local therapy < 2 weeks before the first dose of study intervention;
  5. Non-specific immunomodulatory therapy < 2 weeks before the first dose.
  6. Prior systemic anti-angiogenic therapy
* Prior immune-related AE that led to anti-PD-(L)1 treatment discontinuation, adverse events from prior immunotherapy not improved to Grade 1 before screening, or required treatment with systemic immunosuppressive therapy.
* Prior and concomitant therapy:

  1. therapeutic oral or parenteral anticoagulants or thrombolytic agents < 10 days to the first dose.
  2. chronic antiplatelet therapy <7 days to randomization.
  3. live or attenuated live vaccine < 4 weeks to the first dose.
  4. current high-dose systemic corticosteroids.
  5. prohibited concomitant medication(s) < 21 days to the first dose.
* Breastfeeding participants, participants of childbearing potential, and male participants who are unwilling to follow contraceptive measures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1410 (Estimated)
Dates: Start 2026-01-06 (Actual); Primary Completion 2029-02-27 (Estimated); Study Completion 2032-08-26 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | Approximately 39 months
  Overall survival defined as the time from the date of randomization to the date of death due to any cause.
Progression Free Survival (PFS) assessed by blinded independent central review (BICR) | Approximately 32 months
  Progression-free survival is defined as the time from the date of randomization to the date of the first documentation of objective progressive disease (PD) assessed by BICR per RECIST v1.1, or death due to any cause, whichever occurs first.

SECONDARY OUTCOMES:
Confirmed objective response rate (ORR) using RECIST v1.1 as assessed by BICR | Approximately 32 months
  ORR is defined as the proportion of participants in the analysis population having a best overall response (BOR) of confirmed CR or confirmed PR according to RECIST v1.1 as assessed by BICR.
Progression Free Survival as assessed by Investigator | Approximately 32 months
  Progression Free Survival (PFS) is defined as the time from the date of randomization to the date of the first documentation of objective PD assessed by investigator per RECIST v1.1, or death due to any cause, whichever occurs first.
Confirmed ORR using RECIST v1.1 as assessed by investigator | Approximately 32 months
  ORR is defined as the proportion of participants in the analysis population having a BOR of confirmed CR or confirmed PR according to RECIST v1.1 as assessed by BICR.
Duration of Response (DoR) as assessed by BICR | Approximately 32 months
  The time from the first documentation of objective response (CR or PR that is subsequently confirmed) to the date of the first documentation of PD as determined by BICR assessment per RECIST v1.1, or death due to any cause, whichever occurs first.
Duration of Response (DoR) as assessed by Investigator | Approximately 32 months
  The time from the first documentation of objective response (CR or PR that is subsequently confirmed) to the date of the first documentation of PD as determined by investigator assessment per RECIST v1.1, or death due to any cause, whichever occurs first.
Number of Participants With Adverse Events (AEs) | Through end of study and up to approximately 39 months
  AEs as characterized by type, frequency, intensity as graded by NCI CTCAE version 5.0, timing, seriousness, and relationship to study intervention(s).
Number of Participants With Clinical Laboratory Abnormalities | through end of study and up to approximately 39 months
  Laboratory test abnormalities as characterized by type, frequency, severity (as graded by NCI CTCAE version 5.0) and timing.
Pharmacokinetics (PK): Serum concentrations of PF-08634404 | Through end of study and up to approximately 39 months
  Predose and postdose concentrations of PF-08634404
Incidence of Anti-Drug Antibody (ADA) against PF-08634404. | Through end of study and up to approximately 39 months
Mean scores and Change from baseline in the global health status/quality of life (QoL) and physical function scores on the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30) | Approximately 39 months
  The EORTC QLQ-C30 is a questionnaire for quantitative measure of health-related quality of life pertinent to participants with a broad range of cancers who are participating in international clinical trials.
Time to definitive deterioration (TTdD) in in the global health status/QoL and physical function scores on the EORTC QLQ-C30 | Approximately 39 months
  TTdD is defined as the time from date of randomization to first onset of Patient Reported Outcome (PRO) deterioration without subsequent recovery.
Mean scores and Change from Baseline in dyspnea, cough, and chest pain scores on the EORTC Quality of Life Cancer Questionnaire - Lung Cancer 13 QLQ-LC13 | Approximately 39 months
  EORTC QLQ-LC13 is a lung cancer specific module that serves as an additional 13 item questionnaire to the general EORTC cancer questionnaire, the EORTC QLQ-C30.
TTdD in the dyspnea, cough, and chest pain scores on the EORTC QLQ-LC13 | Approximately 39 months
  TTdD is defined as the time from date of randomization to first onset of Patient Reported Outcome (PRO) deterioration without subsequent recovery.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (17):
- United States (13):
  - Highlands Oncology Group, Springdale, Arkansas
  - Sansum Clinic, California City, California
  - Cancer Care Centers of Brevard, Inc., Melbourne, Florida
  - Mid Florida Hematology and Oncology Center, Orange City, Florida
  - Hope and Healing Cancer Services, New Lenox, Illinois
  - Illinois CancerCare, P.C., Peoria, Illinois
  - Hematology Oncology Associates of Rockland, Nyack, New York
  - Tennessee Cancer Specialists, Knoxville, Tennessee
  - SCRI Oncology Partners, Nashville, Tennessee
  - Texas Oncology - West Texas, El Paso, Texas
  - Texas Oncology - Gulf Coast, Texas City, Texas
  - Texas Oncology - Northeast Texas, Tyler, Texas
  - Northwest Cancer Specialists - Vancouver, Vancouver, Washington
- Icon Cancer Centre Hobart, Hobart, Australia
- National Hospital Organization Kyushu Cancer Center, Fukuoka, Japan
- Puerto Rico (2):
  - Pan American Center for Oncology Trials, LLC- Dorado Office, Dorado
  - BRCR Global Puerto Rico - Hato Rey, San Juan

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C6461001